CLINICAL TRIAL: NCT05012189
Title: Comparative Effectiveness of Baloxavir Versus Oseltamivir for Influenza Outbreak Management in U.S. Nursing Homes
Brief Title: Baloxavir Versus Oseltamivir for Nursing Home Influenza Outbreaks
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Brown University (Other); Case Western Reserve University (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INSI-202107
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Influenza; Influenza, Human; Influenza -Like Illness
Keywords: Antiviral Medication; Influenza; Nursing Home; Influenza Outbreak; Outbreak; Oseltamivir; Baloxavir
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; baloxavir

STUDY DESIGN:
Intervention Model Description: Pragmatic Cluster Randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oseltamivir (Active Comparator): Nursing homes randomized to receive oseltamivir for treatment and chemoprophylaxis for influenza.
  Interventions: Drug: Oseltamivir
- Baloxavir (Experimental): Nursing homes randomized to receive baloxavir for treatment and chemoprophylaxis for influenza.
  Interventions: Drug: Baloxavir

INTERVENTIONS:
Drug: Oseltamivir — Nursing home residents and staff 18 years and older are allocated to receive oseltamivir for treatment and chemoprophylaxis for influenza.
  Arms: Oseltamivir
Drug: Baloxavir — Nursing home residents and staff 18 years and older are allocated to receive baloxavir for treatment and chemoprophylaxis for influenza.
  Arms: Baloxavir

SUMMARY:
Influenza outbreaks are a prevalent event in nursing homes (NHs). We will study baloxavir compared to oseltamivir when used for influenza prophylaxis when facilities identify an index incident case of influenza. This study will help guide nursing home's decision making and demonstrate the effectiveness of a novel antiviral for preventing influenza outbreaks.

DETAILED DESCRIPTION:
A random study sample of about 1000 U.S. nursing homes (NHs), housing approximately 112,000 overall residents and 92,000 over the age of 65 years, of whom 64,500 are long-stay NH residents, will be recruited for the study. Participating facilities will be randomly allocated in a 1:1 ratio to oseltamivir or baloxavir for antiviral treatment and prophylaxis. Primary study data provided by facilities monthly during the influenza season will support primary and secondary endpoints along with administrative claims and public use datasets containing information on facility characteristics.

ELIGIBILITY:
Inclusion Criteria:

- Medicare-certified NHs in any location in the United States with at least 50 long-stay residents 18 years of age or older.

Exclusion Criteria:

* Hospital-based facilities
* Facilities not submitting MDS data

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Total number of ILI cases defined, following the index influenza case identification in nursing homes randomized to baloxavir or oseltamivir | Up to 8 months each influenza season
  To demonstrate the non-inferiority of prophylactic baloxavir vs. oseltamivir to prevent influenza-like illness (ILI) after an index influenza case in nursing homes.

SECONDARY OUTCOMES:
Outbreak duration defined as the time of the first laboratory-confirmed case of influenza to 7 days following the last identified case of influenza-like illness requiring treatment with baloxavir or oseltamivir | Up to 8 months each influenza season
  To determine the difference in total outbreak duration for each outbreak occurring in nursing homes randomized to offer either single-dose baloxavir or oseltamivir for outbreak abatement during the 2021-2022 influenza season.
Facility-level data on antiviral courses of treatment administered from Medication Administration Records | Up to 8 months each influenza season
  To determine the difference in number of courses of treatment of baloxavir or oseltamivir needed for outbreak control in nursing homes randomized to baloxavir or oseltamivir.
Hospitalizations from Minimum Data Set (MDS) 3.0 (interim) and Medicare A claims | Up to 8 months each influenza season
  To determine the difference in respiratory-related hospitalization rates during the 2021-2022 influenza season experienced by long-stay nursing home residents 65 and older living in nursing homes randomized to either baloxavir or oseltamivir.
Mortality from Medicare Vital Status File | Up to 8 months each influenza season
  To determine the differences in long-stay residents' mortality rates in nursing homes randomized to either baloxavir or oseltamivir.

CONTACTS AND LOCATIONS:
Locations (1):
- Insight Therapeutics, LLC, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No